CLINICAL TRIAL: NCT00241917
Title: Cooperative Agreement to Develop, Implement, and Evaluate Viral Hepatitis and Training
Brief Title: A Video-Based HCV Curriculum for Drug Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organization to Achieve Solutions in Substance Abuse (OASIS) (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Diana Sylvestre, MD, OASIS
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: U50/CCU923257; U50/CCU923257
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2008-12-09 (Estimated); Status verified 2008-12

CONDITIONS: Hepatitis C; Opiate Dependence
Keywords: hepatitis C; heroin; populations at risk; testing; vaccination
MeSH Terms: conditions — Hepatitis C; Opioid-Related Disorders | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video (Experimental)
  Interventions: Behavioral: Hepatitis C educational video; Other: Video
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Hepatitis C educational video
  Arms: Video
Other: Video — Prevention education video about hepatitis C
  Arms: Video

SUMMARY:
The investigators hypothesize that a well-designed hepatitis C (HCV)video education curriculum for high-risk drug users will show measurable benefits in improving HCV testing, hepatitis A and B vaccinations, and HCV knowledge, attitudes, and motivations toward transmission behavior change. The investigators will use a 4-part modular video series designed for at-risk drug users, and in this 12 week study will assess its impact on testing/vaccinations as well as knowledge, attitudes, and motivations in methadone-maintained drug users as compared to a usual-care intervention.

DETAILED DESCRIPTION:
Injection drug users are at high risk for contracting hepatitis C (HCV). Very few culturally-specific educational tools have been developed to improve outcomes in this population. We hypothesize that measurable improvements in HCV testing, hepatitis A and B vaccinations, and testable knowledge, attitudes, and motivations may be elicited by such a curriculum.

In this study, we will investigate the impact of a 4-module short video educational series on these measures in in-treatment drug users maintained on methadone. Subjects will be enrolled in 3 sequential cohorts of 150 each: usual care, a 4 weekly sequential video cohort, and a single-session intervention in which the 4 videos are viewed at once. Subjects will undergo written testing for knowledge, attitudes about transmission behaviors, and motivations toward behavior change before the intervention, 4 weeks after the intervention, and 12 weeks after the intervention. Additionally, we will measure and compare the rates of HCV testing and HAV/HBV vaccinations before and at the 12-week time point in all cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Enrolled on methadone maintenance within last 30 days

Exclusion Criteria:

* Unable to provide informed consent
* Not interested in study
* Not able to speak or understand English

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2005-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
HCV testing rates, intervention vs. usual care
HAV vaccination rates, intervention vs. usual care
HBV vaccination rates, intervention vs. usual care

SECONDARY OUTCOMES:
Improvement in knowledge, intervention vs. usual care
Improvement in attitudes toward behavior change, intervention vs. usual care
Improvement in motivation toward behavior change, intervention vs. usual care

CONTACTS AND LOCATIONS:
Overall Officials: Diana L Sylvestre, MD, Principal Investigator — Organization to Achieve Solutions in Substance Abuse (OASIS)
Locations (3):
- United States (3):
  - BAART/Antioch Methadone Clinic, Antioch, California
  - BAART/Richmond Methadone Clinic, Richmond, California
  - BAART/Market Methadone Clinic, San Francisco, California